CLINICAL TRIAL: NCT07234032
Title: A Long-term Open-Label Extension Study of Treprostinil Palmitil Inhalation Powder for Treatment of Pulmonary Hypertension Associated With Interstitial Lung Disease
Brief Title: An Open-Label Extension Study of Treprostinil Palmitil Inhalation Powder (TPIP) in Participants With Pulmonary Hypertension Associated With Interstitial Lung Disease (PH-ILD)
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Insmed Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: INS1009-312; 2025-521769-29-00 (Other: EU CT Number)
Expanded Access: NCT06939647 (Available)
Record Dates: First submitted 2025-11-14; First posted 2025-11-18 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Pulmonary Hypertension; Interstitial Lung Disease
Keywords: pulmonary hypertension, interstitial lung disease
MeSH Terms: conditions — Hypertension, Pulmonary; Lung Diseases, Interstitial

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treprostinil Palmitil Inhalation Powder (TPIP) (Experimental): Participants transitioning from study INS1009-311 (NCT07179380) will undergo an initial double-dummy titration with the stable dose from the lead-in study and either TPIP or placebo for 4 weeks. They will then receive open-label TPIP at a stable maintenance dose with optional escalation (80-1280 micrograms once daily) for the remainder of the 104-week treatment period.
  Interventions: Drug: Treprostinil Palmitil Inhalation Powder; Drug: Placebo

INTERVENTIONS:
Drug: Treprostinil Palmitil Inhalation Powder — Oral inhalation using a capsule-based dry powder.
  Other Names: INS1009
Drug: Placebo — Oral inhalation in initial double-dummy titration period.

SUMMARY:
The primary objective of this study is to evaluate the safety and tolerability of the long-term use of TPIP in participants with PH-ILD from Study INS1009-311 (NCT07179380).

ELIGIBILITY:
Inclusion Criteria

* Participants who have completed the lead-in PH-ILD TPIP Study INS1009-311 (NCT07179380).
* Capable of giving signed informed consent that includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in this protocol.
* Agree not to participate in any other interventional trials or use investigational drugs or devices while participating in the INS1009-312 study.

Exclusion Criteria

* Participants who experienced any adverse events (AEs) evaluated as causally related to TPIP by the Investigator in a lead-in study, which in the opinion of the Investigator, could pose an unreasonable risk of continued treatments for the participant.
* Current use or expected need for pulmonary arterial hypertension (PAH)-approved therapy, including prostacyclin, prostacyclin analogues or other prostacyclin receptor agonists, endothelin receptor antagonists, and/or soluble guanylate cyclase stimulator, or any PH-ILD approved treprostinil therapy. Use of phosphodiesterase 5 inhibitors in line with applicable guidelines is allowed.
* Diagnosis of Pulmonary Hypertension World Health Organisation (WHO) Groups 1, 2, 4, or 5, or subtypes of PH WHO Group 3 other than interstitial lung disease (including combined pulmonary fibrosis and emphysema).
* Evidence of left ventricular failure, heart failure with preserved ejection fraction (HFpEF) or postcapillary PH.
* Known hypersensitivity or contraindication to treprostinil or TPIP or TPIP formulation excipients (eg, mannitol, leucine).

Note: Other protocol-defined inclusion/exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 344 (Estimated)
Dates: Start 2026-04-01 (Estimated); Primary Completion 2031-01-22 (Estimated); Study Completion 2031-01-22 (Estimated)

PRIMARY OUTCOMES:
Number of Participants Who Experienced at Least One Treatment-Emergent Adverse Events (TEAEs) | Up to 108 weeks

SECONDARY OUTCOMES:
Change From Baseline in 6-Minute Walk Distance (6MWD) Measured Post-Dose | Up to 104 weeks
Absolute Change From Baseline in Forced Vital Capacity (FVC) | Up to 104 weeks
Percent Change From Baseline in Forced Vital Capacity (FVC) | Up to 104 weeks
Absolute Change From Baseline in Percent Predicted FVC (FVC% pred) | Up to 104 weeks
Percent Change From Baseline in Percent Predicted FVC (FVC% pred) | Up to 104 weeks
Absolute Change From Baseline in Forced Expiratory Volume in 1 Second (FEV1) | Up to 104 weeks
Percent Change From Baseline in Forced Expiratory Volume in 1 Second (FEV1) | Up to 104 weeks
Absolute Change From Baseline in Percent Predicted FEV1 (FEV1%) | Up to 104 weeks
Percent Change From Baseline in Percent Predicted FEV1 (FEV1%) | Up to 104 weeks
Change From Baseline in the Plasma Concentration of N-Terminal Pro B-Type Natriuretic Peptide (NT-proBNP) | Up to 104 weeks
Annualized Rate of Occurrence of Exacerbations of Interstitial Lung Disease (ILD) | Up to 104 weeks
Percentage of Participants With a Clinical Worsening Events | Up to 104 weeks
Mean Change From Baseline in Living With Pulmonary Fibrosis (L-PF) Domain Score | Up to 104 weeks
Mean Change From Baseline in L-PF Cough Domain Score | Up to 104 weeks
Mean Change From Baseline in L-PF Dyspnea Domain Score | Up to 104 weeks
Mean Change From Baseline in L-PF Impact Domain Score | Up to 104 weeks
Mean Change From Baseline in the EuroQoL- 5 Dimensions (EQ-5D-5L) Index Score | Up to 104 weeks
Mean Change From Baseline in the EQ-5D-5L Visual Analog Scale (VAS) | Up to 104 weeks
Percentage of Participants With Major Morbidity or Mortality Events | Up to 104 weeks

IPD SHARING:
Plan to Share IPD: No